CLINICAL TRIAL: NCT02958059
Title: Effectiveness of Prophylactic Antibiotics to Prevent Post Endoscopic Retrograde Cholangio Pancreatography Bacteremia in Biliary Obstruction Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2015-0596
Record Dates: First submitted 2016-11-01; First posted 2016-11-08 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Biliary Obstructive Disease Such as Choledocholithiasis; Benign Biliary Stricture; Peri-ampullary Cancer; Bile Duct Cancer Resectable; Klatskin Tumor
Keywords: ERCP; prophylaxis; antibiotics; infection; cholangitis
MeSH Terms: conditions — Klatskin Tumor; Infections; Cholangitis | interventions — Cefoxitin; Antibiotic Prophylaxis; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): The intervention group
  Interventions: Biological: Pacetin® (cefoxitin)
- Comparator (Placebo Comparator): The comparator group
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Pacetin® (cefoxitin) — 1~2g of Cefoxitin (2nd generation cephalosporin) is administered to patients 30 minutes Before ERCP procedure. Cefoxitin is mixed with 10ml of normal saline. Patients and caregivers can not distinguish antibiotics and placebo by naked eye.
  Other Names: Antibiotic prophylaxis
  Arms: Treatment
Biological: Placebo — 10ml of normal saline is injected to patients as placebo. Patients and caregivers can not distinguish antibiotics and placebo by naked eye.
  Other Names: normal saline
  Arms: Comparator

SUMMARY:
Endoscopic retrograde cholangio-pancreatography (ERCP) is advanced endoscopic technique that allows minimally invasive management of biliary and pancreatic disorders. However, the incidence of infectious complication of ERCP is considerable. Transient blood stream infection after ERCP has been reported in a high ratio, up to 27% and post-ERCP infection accounts for about 10% of the major complications associated with mortality.

Although prophylactic use of antibiotics is generally not recommend in all cases, debates about the prophylactic use of antibiotics continues and prophylactic use of antibiotics is recommend in case of ERCP that incomplete biliary drainage is expected.

In this study, researchers will use prophylactic antibiotics in patients with biliary obstruction who have high-risk of post-ERCP bacteremia. Antibiotics regimen is selected based on the data of our institution, and administered to patients before ERCP procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biliary obstructive disease (Benign or Malignant)
* 19 year-old and older than 19 year-old

Exclusion Criteria:

* Younger than 19 year-old
* Patients with leukocytosis (WBC ≥ 11,000/mm3)
* Body temperature ≥ 38 °C within 72 hours before ERCP
* History of antibiotics administration due to cholangitis, cholecystitis or sepsis within 72 hours before ERCP
* Pregnancy women
* Patients with allergy to beta-lactam

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Rate of complication that related with infection. | within 10 days

SECONDARY OUTCOMES:
Rate of post-ERCP cholangitis | within 10 days
Grade of post-ERCP infectious complication | within 10 days
  Grade of post-ERCP infectious complications based upon a consensus definition Mild : >38°C for 24-48 hr / Moderate : Febrile or septic illness requiring more than 3 days of hospital treatment or endoscopic or percutaneous intervention / Severe : Septic shock or surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university of medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leem G, Sung MJ, Park JH, Kim SJ, Jo JH, Lee HS, Ku NS, Park JY, Bang S, Park SW, Song SY, Chung MJ. Randomized Trial of Prophylactic Antibiotics for Endoscopic Retrograde Cholangiopancreatography in Patients With Biliary Obstruction. Am J Gastroenterol. 2024 Jan 1;119(1):183-190. doi: 10.14309/ajg.0000000000002495. Epub 2023 Sep 15. PMID 37713527